CLINICAL TRIAL: NCT06241248
Title: Evaluation of the Performance of a New Rapid Bacteremia Test in the Intensive Care Patient
Acronym: OCEANIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/28
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Sepsis
Keywords: Intensive Care; Blood culture; Bacteremia; Rapid Diagnostic Tests; Antimicrobial resistance
MeSH Terms: conditions — Sepsis; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood bacterial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ocean Test: The OCEAN Dx tests for the diagnosis of sepsis will be performed on 9 milliliters of blood collected at the patient's bedside.The sample will be collected at the same time as the blood cultures are taken. The blood tubes will then be transported to OCEAN Dx laboratories.
  Interventions: Diagnostic Test: Rapid sepsis diagnostic test

INTERVENTIONS:
Diagnostic Test: Rapid sepsis diagnostic test — The different stages of the OCEAN Dx whole blood bacterial identification test. Identification is carried out using 9 ml of whole blood taken at the patient's bedside, and is provided after comparing the DNA sequence of the bacteria with a database. The rapid sepsis diagnostic test developed by OCEAN Dx can identify the bacteria responsible for the infection in just 4 hours at present, and soon in 3 hours. Subject to future innovations, it will probably even be possible to obtain a positive result for the presence of bacteria in the patient's sample in just 2 hours.

SUMMARY:
Sepsis is a serious health problem with a very high mortality in the ICU. The most important treatment for sepsis is the fastest possible antibiotic therapy. The identification of the pathogen responsible for sepsis is essential to propose an appropriate antibiotic treatment. However, the diagnosis of bacteremia by blood culture requires an average delay of 48 to 72 hours. The new test proposed by OCEAN Dx makes it possible to identify a bacteremia in a few hours. The main objective of the study is to evaluate the performance of the rapid identification test for bacteremia proposed by OCEAN Dx compared to a classic diagnostic strategy using blood cultures.

DETAILED DESCRIPTION:
Sepsis is a worldwide problem. The World Health Organization estimates that around 49 million people suffer from sepsis each year. It is responsible for an unacceptable number of deaths, estimated at around 11 million. The severity of sepsis is not only related to the infection itself, but often to a too late diagnosis and an important heterogeneity in the management of patients. The identification of the pathogen responsible for sepsis is currently based on the positivity of bacteriological samples, particularly blood cultures. However, the diagnosis of bacteremia by blood cultures requires an average delay of 48 to 72 hours, which is not conducive to rapid adaptation of antibiotic therapy. The test proposed by OCEAN Dx offers the identification of a bacteremia in a few hours thanks to the recognition of the bacterial DNA in the patient's blood. The main objective of the study is to evaluate the performance of the rapid identification test for bacteremia offered by OCEAN Dx in comparison with a classical diagnostic strategy using blood cultures.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age admitted to an intensive care unit (ICU) with a suspected or documented infection requiring blood cultures.

Exclusion Criteria:

* Patient under 18 years of age
* Pregnant or breastfeeding woman
* Patient of legal age, under guardianship or deprived of liberty
* Not affiliated to a social security regime or not benefiting from such a regime.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to an intensive care unit (ICU) with a suspected or documented infection requiring blood cultures
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Comparison between OCEAN test and gold standard | 1 month after inclusion day
  Agreement between the OCEAN Dx test results and blood cultures, gold standard of bacteriemia identification.

SECONDARY OUTCOMES:
Positivity rate | 1 month after inclusion day
  The positivity rate of the OCEAN Dx test and blood cultures
Delay of positivity | 1 month after inclusion day
  Time to positivity of the OCEAN Dx test and blood cultures
Impact of Ocean test on antibiotic therapy adaptation. | 1 month after inclusion day
  Cost of prescribed antibiotics and theoretical antibiotics after de-escalation according to the identification of germs by blood cultures and the OCEAN Dx test

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Haut-Lévêque, Pessac, France

IPD SHARING:
Plan to Share IPD: No